CLINICAL TRIAL: NCT04211779
Title: The Effect of Anodal Transcranial Direct Current Stimulation Combined With Aerobic Exercise on Performance in Healthy Individuals
Brief Title: a-tDCS Combined With Aerobic Exercise in Healthy Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 09.2019.669
Record Dates: First submitted 2019-12-19; First posted 2019-12-26 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2019-12

CONDITIONS: Healthy
Keywords: Transcranial Direct Current Stimulation; Aerobic Exercise; Performance
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Real tDCS and Exercise (Experimental): tDCS (tDCS - TCT Research Limited, Hong Kong) / Exercise Group in which will receive the active intervention of aerobic exercise training and active tDCS intervention at the same time.
  Interventions: Device: Real tDCS; Other: Exercise
- Sham tDCS and Exercise (Sham Comparator): Sham tDCS (tDCS - TCT Research Limited, Hong Kong) / Exercise Group in which will receive the active intervention of aerobic exercise training and sham tDCS intervention at the same time.
  Interventions: Device: Sham tDCS; Other: Exercise
- Exercise (Other): Exercise group in which will receive the active intervention of aerobic exercise training no tDCS intervention.
  Interventions: Other: Exercise

INTERVENTIONS:
Device: Real tDCS — Real tDCS (TCT Research Limited, Hong Kong); 3 times a week on alternate days for consecutive 6 weeks. The active session of tDCS will consist in applying anodal stimulation over left M1 (C3 according to the 10-20 international EEG placement) and the cathodal stimulation over right supraorbital area (Fp2 according to the 10-20 international EEG placement), and to inject 2 mA for 20 minutes through sponge electrodes (35 cm²) placed on the scalp.
  Arms: Real tDCS and Exercise
Device: Sham tDCS — Sham current (TCT Research Limited, Hong Kong); 3 times a week on alternate days for consecutive 6 weeks. The sham tDCS will use the same montage and device but direct current will only be injected for 30 seconds, with a ramp-up and ramp-down 15 seconds period, to mimic the somatosensory effects of active tDCS.
  Arms: Sham tDCS and Exercise
Other: Exercise — The Exercise intervention will include only aerobic exercise 3 times a week on alternate days for consecutive 6 weeks. The program will last 20 minutes.

SUMMARY:
The purpose of this study is to assess the effects on the exercise performance of anodal transcranial direct current stimulation combined with aerobic exercise in healthy individuals.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation method that has become increasingly popular in recent years. tDCS shows promising improvements for the motor performance of healthy individuals as well as pathological conditions. Moreover, it is frequently preferred because of its safety advantage, high tolerability as well as being cheap, portable and easily applicable.

Studies have shown that tDCS can modulate the excitability of both cortical and subcortical brain regions. In recent years, there have been scientific studies investigating the effects of tDCS on improving physical performance in healthy individuals, but these studies are limited in number, their results are conflicted and as far as the investigators know there is no study that combines tDCS with exercise.

Moreover, although the mechanisms of tDCS on physical performance are largely unknown, some tDCS devices are open to public usage and a large number of professional athletes have reported using tDCS during their training programs. Therefore, studies are needed to demonstrate the effects of tDCS which combined with exercise on performance.

The aim of this study was to investigate the effects of anodal transcranial direct current stimulation combined with aerobic exercise on physical performance in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject
* No use of any ergogenic substance in one year
* No history of active exercise training in last 6 months

Exclusion Criteria:

* Pacemaker
* Intracerebral metallic implant
* Using dietary supplementation or medication potentially affecting the CNS
* Musculoskeletal injury within the past 6 weeks
* Lower extremity pain above 3 or more according to numeric pain scale
* History of epilepsy or convulsive crisis

Ages: 20 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-10-29 (Estimated); Study Completion 2021-12-29 (Estimated)

PRIMARY OUTCOMES:
Effect of tDCS combined with aerobic exercise on exercise performance in healthy individuals. | 2 months
  The performance will be evaluated by measuring the maximal consumption of oxygen (VO2max). VO2max will be assessed continuously during the time to exhaustion trial using a gas analyzer
Effect of tDCS combined with aerobic exercise on ratings of perceived exertion (RPE) in healthy individuals. | 2 months
  RPE will be assessed continuously (every 3 minutes) during the time to exhaustion trial using the Borg rating of perceived exertion scale (RPE scale). The Borg RPE scale is a quantitative measure of perceived exertion during physical activity. The scale starts with "no feeling of exertion," which rates a 6, and ends with "very, very hard," which rates a 20. Moderate activities register 11 to 14 on the Borg scale ("fairly light" to "somewhat hard"), while vigorous activities usually rate a 15 or higher ("hard" to "very, very hard").

SECONDARY OUTCOMES:
Effect of tDCS combined with aerobic exercise on isokinetic muscle strength in healthy individuals. | 2 months
  The isokinetic muscle strength of knee extensors of the dominant leg will be evaluated by using Biodex System 3 isokinetic dynamometer (Biodex Medical Systems, Shirley, NY, USA)

OTHER OUTCOMES:
Changes in SF-36 questionnaire of quality of life | 2 months
  This questionnaire evaluates different aspects of individual life such as Vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Through different questions, a score is generated for each subscale where zero represents the worst quality of life and 100 the best quality of life.
Changes in Cognitive Test Battery | 2 months
  An n-back cognitive test will be conducted for assessing the working memory.

CONTACTS AND LOCATIONS:
Overall Officials: Mine Gülden Polat, PhD, Study Director — Marmara University; Lütfü Hanoğlu, PhD, Study Chair — Medipol University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No